CLINICAL TRIAL: NCT04427020
Title: Changes in Amino Acid Absorption After Adding a Probiotic to an Acute Protein Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-20-15
Record Dates: First submitted 2020-06-01; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Amino Acid Absorption
MeSH Terms: interventions — Milk Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Protein and probiotics were delivered separately. Upon arrival a faculty member (who was not an investigator) blinded both the protein and probiotic samples and kept the code sealed in an envelope until all statistical analysis was complete. Once all data collection, data entry, and statistical analysis was completely finished, the study code was broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk Protein + Probiotic (Experimental): 25 gram dose of milk protein concentrate with bacillus coagulans GBI-30, 6086
  Interventions: Dietary Supplement: Milk protein + GBI-30
- Milk Protein (Active Comparator): 25 gram dose of milk protein concentrate
  Interventions: Dietary Supplement: Milk protein

INTERVENTIONS:
Dietary Supplement: Milk protein + GBI-30 — Both conditions matched flavor, color, and serving size
  Arms: Milk Protein + Probiotic
Dietary Supplement: Milk protein — Both conditions matched flavor, color, and serving size
  Arms: Milk Protein

SUMMARY:
The purpose of this study is to examine the pharmacokinetic pattern of amino acid absorption after a two-week pattern of milk protein supplementation with and without the addition of Bacillus coagulans GBI-30, 6086.

DETAILED DESCRIPTION:
The study will be conducted using a randomized, double-blind, crossover study design. 30 healthy men and women between the ages of 18 - 55 years of age will be recruited to participate in this study. Prior to beginning the study, all participants will sign an IRB-approved informed consent document and complete a healthy history questionnaire to determine study eligibility. Two supplementation protocols that each span two weeks will be completed and separated with a washout period of three weeks. For each study visit, all participants will report to the laboratory between 0600 - 1000 hours after observing an 8 - 10-hour fast. For two weeks prior to each study visit, participants will be assigned in a randomized, double-blind, crossover fashion to ingest a single daily 25-gram dose of a milk protein concentrate or a similar dose of milk protein concentrate plus bacillus coagulans GBI-30, 6086. Upon arrival for each study visit, participants will have their resting heart rate, blood pressure, body mass, height, and body composition measured using bioelectrical impedance analysis (BIA). Upon ingestion of their final assigned supplementation dose, standard multiple sample phlebotomy approaches will used to collect approximately 10mL of venous blood from a forearm vein before (0 min), 30, 60, 90, 120, 180, and 240 minutes after ingestion of their final assigned supplementation dose for that period in the study protocol. Participants will be provided 200 mL of cold water to ingest after each blood collection. Upon processing, all blood samples will be stored at -80 C. All samples will o be discarded according to Institutional Review Board-stipulated guidelines. Study participants will be provided an additional two-week supply of the alternative treatment to begin after observing a three-week washout. After two weeks of supplementation, study participants will return to the laboratory for their remaining testing visit. All subsequent study visits will be completed in a randomized fashion to minimize any order effects from testing.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be between the ages of 18-55 years.
* Participants will be healthy and free of disease as determined by evaluation of a medical history.
* Completing at least 30 minutes of moderate exercise three days per week

Exclusion Criteria:

* Those individuals less than 18 and greater than 55 years of age will be excluded.
* Any individual who is currently being treated for or diagnosed with a cardiac disorder or disease
* Any individual who is currently being treated for or diagnosed with a respiratory disorder or disease
* Any individual who is currently being treated for or diagnosed with a circulatory disorder or disease
* Any individual who is currently being treated for or diagnosed with a musculoskeletal disorder or disease
* Any individual who is currently being treated for or diagnosed with a metabolic disorder or disease
* Any individual who is currently being treated for or diagnosed with obesity (defined as body mass index > 30 kg/m and body fat greater than 30%)
* Any individual who is currently being treated for or diagnosed with an immune or autoimmune disorder or disease
* Any individual who is currently being treated for or diagnosed with a psychiatric disorder or disease
* Any individual who is currently being treated for or diagnosed with a hematological disorder or disease
* Any individual who is currently being treated for or diagnosed with a neurological disorder or disease
* Any individual who is currently being treated for or diagnosed with an endocrinological disorder or disease
* Participants who are determined to not be weight stable defined as measured body mass deviating by 2% or more.
* Participants who do not or are not willing to abstain from alcohol, nicotine, and caffeine for 12 hours prior to each visit will be excluded
* Participants who do not or are not willing to abstain from exercise for 12 hours prior to each visit will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Rate of amino acid absorption | seven weeks
  We intend to determine if the addition of a probiotic to milk protein ingestion changes the rate (in minutes) to which amino acids are absorbed into our bloodstream.
Concentration of amino acid absorption | seven weeks
  We intend to determine if the addition of a probiotic to milk protein ingestion changes the extent (concentration in millimoles/Liter) to which amino acids are absorbed into our bloodstream.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Kerksick, PhD, Study Director — Laboratory Director
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
All approved unidentified study data inside the laboratory will be saved within a research repository bank for future research questions. Otherwise, participant data will be destroyed after three years of study completion to maintain IRB compliance.

REFERENCES:
- [Derived] Stecker RA, Moon JM, Russo TJ, Ratliff KM, Mumford PW, Jager R, Purpura M, Kerksick CM. Bacillus coagulans GBI-30, 6086 improves amino acid absorption from milk protein. Nutr Metab (Lond). 2020 Oct 23;17:93. doi: 10.1186/s12986-020-00515-2. eCollection 2020. PMID 33110439